CLINICAL TRIAL: NCT03611621
Title: A Prospective Observational, Long Term Follow up Study of Patients Treated With Imlifidase Prior to Kidney Transplantation
Brief Title: A Follow up Study of Patients Treated With Imlifidase Prior to Kidney Transplantation
Status: Completed | Type: Observational
Sponsor: Hansa Biopharma AB (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-HMedIdeS-14
Record Dates: First submitted 2018-07-05; First posted 2018-08-02 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Kidney Transplant Failure and Rejection
MeSH Terms: conditions — Rejection, Psychology | interventions — Mac-1-like protein, Streptococcus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (storage time: maximum 2 years after completion of the study report according to local regulations)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Imlifidase — This is a five year, long-term follow up, observational study. The study will primarily determine the time of graft survival in subjects who have received imlifidase prior to kidney transplantation. Subjects who have participated, or are currently participating, in the imlifidase kidney transplantation studies (called feeder studies) 13-HMedIdeS-02, 13-HMedIdeS-03, 14-HMedIdeS- 04 and 15-HMedIdeS-06 will be included. The subjects will attend 4 follow up visits, 1, 2, 3 and 5 years after imlifidase administration.
  Other Names: IdeS, HMED-IdeS

SUMMARY:
The rationale for the current protocol is to collect data from extended follow up in subjects that have received a kidney transplant following imlifidase dosing to provide a better understanding regarding the long-term outcome for these subjects. Data of parameters such as patient and graft survival, comorbidity, treatment of graft rejection episodes and quality of life as well as anti-drug antibody levels will be collected.

This prospective, observational follow up study of subjects who have received imlifidase prior to kidney transplantation will provide important data to future prescribers and patients of the potential long-term benefits of imlifidase mediated transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent obtained before any study-related procedures
* Previous dosing with imlifidase followed by kidney transplantation and participation in one of the following clinical studies: 13-HMedIdeS-02, 13-HMedIdeS-03, 14-HMedIdeS-04 or 15-HMedIdeS-06

Exclusion Criteria:

* Individuals deemed unable to comply with the protocol
* Inability by the judgment of the investigator to participate in the study for other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects that have participated, or are currently participating, in the imlifidase kidney transplantation studies; 13-HMedIdeS-02, 13-HMedIdeS-03, 14-HMedIdeS-04 and 15-HMedIdeS-06 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Director — Hansa Biopharma AB
Locations (6):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - New York University School of Medicine, New York, New York
- Necker Hospital, Paris, France
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Long-term follow-up of patients participating in the imlifidase kidney transplantation studies (feeder studies) 13-HMedIdeS-02, 13-HMedIdeS-03, 14-HMedIdeS-04 and 15-HMedIdeS-06. The patients attend 4 follow up visits, 1, 2, 3 and 5 years after imlifidase administration. Up to 46 patients could be included depending on patients' willingness to participate in the trial.
Pre-assignment Details: Data from patients who died (n=3) or had lost their graft (n=3) after the end of the feeder study but prior to being enrolled in the current trial, were included in the data analysis after ethics permission i.e. data from 37 patients was analyzed.
Groups:
- Imlifidase: All patients
Period: Overall Study
Arm/Group | Imlifidase
Started | 37 (Data from patients who died (n=3) or had lost their graft (n=3) after the end of the feeder study but prior to being enrolled in the current trial, were included in the data analysis after ethics permission.)
Completed | 30
Not Completed | 7
Not completed — Graft loss | 3
Not completed — Death | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Baseline data at time of enrollment in feeder studies
Arm/Group | Imlifidase
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 27
  Race: Asian | 4
  Race: Black or African American | 4
  Race: Other | 2
Region of Enrollment [Number; unit: participants]
  Sweden | 13
  United States | 22
  France | 2
Height [Mean (Standard Deviation); unit: cm] | 171.4 (10.1)
Weight [Mean (Standard Deviation); unit: kg] | 72.2 (15.1)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 24.2 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Graft Survival in Subjects Who Have Undergone Kidney Transplantation After Imlifidase Administration.
Description: The primary endpoint of this study is to determine overall graft survival, defined as time from transplantation to graft loss.
Time Frame: 5 years after first dose of imlifidase (in the feeder study)
Population: The primary endpoint, overall graft survival, was analyzed by the Kaplan-Meier survival method and presented with 95% confidence limits. The following events were censored at the time of occurrence: withdrawal from the trial without graft loss, death not caused by graft loss, and end of trial without graft loss.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Imlifidase
Number analyzed (Participants) | 37
percentage | 91 [75 to 97]

2. Secondary Outcome: Evaluation of Long-term Clinical Outcomes of Transplanted Subjects Treated With Imlifidase in Terms of Patient Survival.
Description: Overall patient survival defined as time from transplantation to death for any cause
Time Frame: 5 years after first dose of imlifidase (in the feeder study)
Population: The overall patient survival was analyzed by the Kaplan-Meier survival method and presented with 95% confidence limits. The following events were censored: withdrawal from the trial while alive, and end of trial while alive
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Imlifidase
Number analyzed (Participants) | 37
percentage | 92 [77 to 97]

3. Secondary Outcome: Evaluation of Long-term Clinical Outcomes of Transplanted Subjects Treated With Imlifidase in Terms of Kidney Function (Estimated Glomerular Filtration Rate (eGFR)).
Description: Kidney function as evaluated by estimated glomerular filtration rate (eGFR). eGFR was calculated according to the Modification of Diet in Renal Disease (MDRD) equation.
Time Frame: 5 years after first dose of imlifidase (in the feeder study)
Population: Patients with a visit/assessment at year 5
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | Imlifidase
Number analyzed (Participants) | 30
mL/min/1.73m2 | 50.74 (19.38)

4. Secondary Outcome: Evaluation of Long-term Clinical Outcomes of Transplanted Subjects Treated With Imlifidase in Terms of Kidney Function (Plasma (P)-Creatinine).
Description: Kidney function as evaluated by analysis of plasma (P)-creatinine
Time Frame: 5 years after first dose of imlifidase (in the feeder study)
Population: Patients with a visit/assessment at year 5
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Imlifidase
Number analyzed (Participants) | 30
μmol/L | 141.3 (69.9)

5. Secondary Outcome: Evaluation of Long-term Clinical Outcomes of Transplanted Subjects Treated With Imlifidase in Terms of Kidney Function (Proteinuria).
Description: Kidney function as evaluated by proteinuria by dipstick analysis
Time Frame: 5 years after first dose of imlifidase (in the feeder study)
Population: Patients with a visit/assessment at year 5
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase
Number analyzed (Participants) | 30
Participants
  Positive | 14
  Negative | 13
  Not done | 3

6. Secondary Outcome: Evaluation of Long-term Clinical Outcomes of Transplanted Subjects Treated With Imlifidase in Terms of Number of Graft Rejection Episodes.
Description: Recording of occurrence of graft rejection episodes classified by Banff criteria (Haas et al 2018).
  The following criteria had to be fulfilled by the rejection episode to constitute an antibody-mediated rejection (AMR):
  * a biopsy was taken at the time of the graft rejection episode
  * histological evidence of an AMR was reported in the pathology report
  * presence of detectable levels of donor specific antibodies (DSAs) and/or evidence of antibody-mediated morphological changes in the kidney transplant at the time of the biopsy
Time Frame: 5 years after first dose of imlifidase (in the feeder study)
Population: Patients with a visit/assessment at year 5. Note: number of patients with suspected acute rejection episodes up until year 5. One (1) biopsy confirmed rejection episode (AMR) was reported for 1 patient approx. 9 months after transplantation. One (1) biopsy confirmed rejection episode reported in the current trial occurred in the feeder trial. Five (5) rejection episodes were not confirmed by biopsy.
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase
Number analyzed (Participants) | 30
Participants
  0 suspected acute rejection episodes | 23
  1 suspected acute rejection episode | 7

7. Secondary Outcome: Evaluation of Long-term Clinical Outcomes of Transplanted Subjects Treated With Imlifidase in Terms of Treatment of Graft Rejection Episodes.
Description: Recording of graft rejection episodes treatments (e.g. dialysis, plasmapheresis and medications).
Time Frame: 5 years after first dose of imlifidase (in the feeder study)
Population: Patients with a visit/assessment at year 5. Any medication (e.g. Intravenous immunoglobulin [IVIg]) given for graft rejection episodes
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase
Number analyzed (Participants) | 30
Participants | 2

8. Secondary Outcome: Evaluation of Long-term Clinical Outcomes of Transplanted Subjects Treated With Imlifidase in Terms of Comorbidities.
Description: Recording of comorbidities up until year 5 after treatment with imlifidase
Time Frame: 5 years after first dose of imlifidase (in the feeder study)
Population: All patients with a comorbidity reported. Note: any single patient could have more than one comorbidity reported.
Measure: Number; unit: participants with comorbidity
Arm/Group | Imlifidase
Number analyzed (Participants) | 18
participants with comorbidity
  urinary tract infection | 9
  nasopharyngitis | 3
  pyelonephritis | 3
  upper respiratory infection | 4
  Covid-19 infection | 4
  urosepsis | 2
  sepsis | 2
  pneumonia | 2
  diabetes mellitus | 4

9. Secondary Outcome: Evaluation of Long-term Clinical Outcomes of Transplanted Subjects Treated With Imlifidase in Terms of Treatments of Comorbidities.
Description: Recording of concomitant immunosuppressive medication
Time Frame: 5 years after first dose of imlifidase (in the feeder study). Note: concomitant immunosuppressive medication up until year 5
Population: Immunosuppressive medications were recorded for 30 of the 31 patients enrolled
Measure: Number; unit: participants
Arm/Group | Imlifidase
Number analyzed (Participants) | 30
participants
  Tacrolimus | 29
  Belatacept | 1
  Mycophenolate | 30
  Prednisone/prednisolone | 30

10. Secondary Outcome: Assessment of Safety Laboratory Testing in Terms of Hematology (Hb)
Description: Blood samples were analyzed for hemoglobulin (Hb)
Time Frame: 5 years after first dose of imlifidase (in the feeder study)
Population: All patients with a visit/assessment at year 5
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Imlifidase
Number analyzed (Participants) | 30
g/L | 121.5 (35.3)

11. Secondary Outcome: Assessment of Safety Laboratory Testing in Terms of Hematology (Differential Analysis of Leucocytes)
Description: Differential analysis of leucocytes was done in blood samples
Time Frame: 5 years after first dose of imlifidase (in the feeder study)
Population: All patients with a visit/assessment at year 5. Note: not all patients had an assessment reported at year 5.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Imlifidase
Number analyzed (Participants) | 30
percentage
  Basophils/Leucocytes: number analyzed (Participants) | 9
  Basophils/Leucocytes | 0.4 (0.19)
  Eosinophils/Leucocytes: number analyzed (Participants) | 8
  Eosinophils/Leucocytes | 1.3 (0.80)
  Lymphocytes/Leucocytes: number analyzed (Participants) | 9
  Lymphocytes/Leucocytes | 20.3 (8.71)
  Monocytes/Leucocytes: number analyzed (Participants) | 9
  Monocytes/Leucocytes | 9.9 (4.87)
  Neutrophils/Leucocytes: number analyzed (Participants) | 8
  Neutrophils/Leucocytes | 56.7 (22.76)

12. Secondary Outcome: Assessment of Safety Laboratory Testing in Terms of Hematology (Thrombocytes)
Description: Blood samples were analyzed for thrombocytes
Time Frame: 5 years after first dose of imlifidase (in the feeder study)
Population: All patients with a visit/assessment at year 5
Measure: Mean (Standard Deviation); unit: 10^9 thrombocytes/L
Arm/Group | Imlifidase
Number analyzed (Participants) | 30
10^9 thrombocytes/L | 225 (65.8)

13. Secondary Outcome: Assessment of Safety Laboratory Testing in Terms of Total Immunoglobulin G (IgG)
Description: Blood samples were analyzed for total IgG levels.
Time Frame: 5 years after first dose of imlifidase (in the feeder study)
Population: All patients with a visit/assessment at year 5.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Imlifidase
Number analyzed (Participants) | 22
g/L | 10.04 (3.96)

14. Secondary Outcome: Assessment of Donor Specific Antibodies (DSA)
Description: DSA levels in blood samples were analyzed by Single Antigen Bead-Human Leukocyte Antigen (SAB-HLA) analysis
Time Frame: 5 years after first dose of imlifidase (in the feeder study)
Population: All patients with a visit/assessment at year 5
Measure: Mean (Standard Deviation); unit: Mean fluorescence intensity (MFI)
Arm/Group | Imlifidase
Number analyzed (Participants) | 20
Mean fluorescence intensity (MFI) | 803 (2038)

15. Secondary Outcome: Assessment of the Presence of BK Virus
Description: Blood samples were analyzed for antibodies towards BK virus
Time Frame: 5 years after first dose of imlifidase (in the feeder study)
Population: All patients with a visit/assessment at year 5
Measure: Number; unit: participants
Arm/Group | Imlifidase
Number analyzed (Participants) | 28
participants
  Presence of BK virus | 0
  No presence of BK virus | 28

16. Secondary Outcome: Assessment of the Immunogenicity of Imlifidase
Description: Serum samples were analyzed for anti-drug antibody (ADA) levels using an ImmunoCAP assay.
Time Frame: 5 years after first dose of imlifidase (in the feeder study)
Population: All patients with a visit/assessment at year 5
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Imlifidase
Number analyzed (Participants) | 20
mg/L | 26.70 (25.42)

17. Secondary Outcome: Evaluation of Long-term Clinical Outcomes of Transplanted Subjects Treated With Imlifidase in Terms of Quality of Life (EQ-5D-5L).
Description: Health related quality of life (HR-QoL) as evaluated by patient questionnaires EQ-5D-5 levels (5L)
  EQ-5D-5L index score values were calculated from individual health profiles by using the corresponding EQ-5D-5L crosswalk value set per country where a higher value correspond to better health. Index score value ranges per country: USA [-0.109 - 1.000], France [-0.530 - 1.000], Denmark [-0.624 - 1.000], since no index score values exist for Sweden, values for Denmark were used for patients from Sweden.
  The visual analogue scale (EQ VAS) score was graded from 0 (the worst imaginable health) to 100 (the best imaginable health), where higher scores correspond to better health.
Time Frame: 5 years after first dose of imlifidase (in the feeder study)
Population: All patients with a visit/assessment at year 5
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Imlifidase
Number analyzed (Participants) | 27
score on a scale
  EQ VAS score | 80.00 [60.00 to 100.00]
  EQ-5D-5L index value USA: number analyzed (Participants) | 13
  EQ-5D-5L index value USA | 0.86 [0.55 to 1.00]
  EQ-5D-5L index value France: number analyzed (Participants) | 2
  EQ-5D-5L index value France | 1.00 [1.00 to 1.00]
  EQ-5D-5L index value Sweden: number analyzed (Participants) | 12
  EQ-5D-5L index value Sweden | 0.79 [0.62 to 1.00]

18. Secondary Outcome: Evaluation of Long-term Clinical Outcomes of Transplanted Subjects Treated With Imlifidase in Terms of Quality of Life (KDQOL-SF).
Description: Health related quality of life (HR-QoL) as evaluated by patient questionnaires Kidney Disease Quality of Life Questionnaire-short form (KDQOL-SF)
  Scores of different subscales were calculated according to the KDQOL-36 scoring program. The scale range for each subscale is 0 to 100, with higher scores indicating better quality of life.
Time Frame: 5 years after first dose of imlifidase (in the feeder study)
Population: All patients with a visit/assessment at year 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Imlifidase
Number analyzed (Participants) | 27
score on a scale
  Burden of kidney disease | 79.4 (22.1)
  Effects of kidney disease | 89.0 (9.9)
  Overall health rating | 76.0 (13.4)
  Cognitive function | 86.9 (18.0)
  Physical functioning | 86.0 (17.6)
  Work status | 74.0 (40.1)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) related to trial procedures or to clinically significant safety laboratory values were recorded from time of informed consent to end of trial, up to 4y and 6m. AEs were not collected for the 6 patients that had lost their graft (n=3) or who died (n=3) after the end of the feeder trials, since these patients were not actively enrolled in the current trial. In the feeder trials AEs were recorded for each patient from time of informed consent to end of trial, up to 6 months.
Description: Only AEs related to trial procedures or to clinically significant safety laboratory values were to be reported in the trial. No AEs or serious adverse events (SAEs) were reported in the trial however 3 graft losses (1 due to infection,1 immunosuppression non-adherence, 1 rejection/loss of function) and 3 deaths (1 circulatory arrest, 1 pseudomonas bacteremia, 1 unknown reason) occurred after the completion of the feeder trials. None of these patients were actively enrolled in the current trial.
Groups:
- Imlifidase: All patients
  Note: AEs were not collected for the patients that lost their graft (n=3) or who died (n=3) after the end of the feeder trials, since they were not actively enrolled in the current trial.
Arm/Group | Imlifidase
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT03611621/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT03611621/SAP_001.pdf